CLINICAL TRIAL: NCT05554003
Title: An Italian Multicenter Phase II Trial of Metronomic Temozolomide in Unfit Patients With Advanced Neuroendocrine Neoplasms (NENs): MeTe Study
Brief Title: Metronomic Temozolomide in Unfit NENs Patients Metronomic Temozolomide in Unfit Patients With Advanced Neuroendocrine Neoplasms (NENs): MeTe Study
Acronym: MeTe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO1411
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Neuroendocrine Tumors; Frailty; Chemotherapy Effect
Keywords: Temozolomide; Neuroendocrine tumors; NETs; NENs; Unfit; Chemotherapy; Metronomic; Advanced; Phase II; Open label
MeSH Terms: conditions — Neuroendocrine Tumors; Frailty | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metronomic Temozolomide (Experimental): Metronomic Temozolomide in unfit patients with advanced neuroendocrine neoplasms (NENs) Dosage and schedule: 60 mg/die continuosly
  Interventions: Drug: Temozolomide capsule

INTERVENTIONS:
Drug: Temozolomide capsule — Metronomic temozolomide 60 mg/die continuously

SUMMARY:
Study design and rationale: Neuroendocrine neoplasms (NENs ) represent a heterogeneous group of malignancies, which differ in terms of behavio r and prognosis. Most of t hem are advanced at diagnosis t herefore systemic treatment is proposed. While over the last years many advanced have been made especially in terms of molecular targeted therapies (MTA) like everolimus and sunitinib, chemotherapy i n NENs still represents a controversial question. Temozolomide has been reported to be active alone or in combination with other drugs in neuroendocrine neoplasms (NENs) from different origin. So far there is not universal agreement on the right setting an d way of administration of this therapy. Objective: This is a multicentric phase II prospective interventional study to evaluate the clinical features of patients, who are judged unfit for systemic treatments, consecutively treated with a metronomic Temozolomide chemotherapy schedule in Italian centers with expertise in NEN and to explore also the methylation status of O6-methylguanine-DNA-methyltransferase (MGMT) and the polymorphism of thymidylate synthase (TS) by pyrosequencing in those patients of which tissues were available. This study will allow a better understanding of the role of metronomic temozolomide chemotherapy in NENs patients and help clinicians in answering some of the outstanding questions on their management. Method: Prospective analysis of clinical data of patients unfit for chemotherapy consecutively treated with metronomic temozolomide regimen in Italian centers with expertise in clinical and research NEN activity, for one year from the start of the accrual. Planning of study: Data from NENs patients of any age treated at these centers will be retrieved by searching the hospital information system and analysed. Eligible study population: Patients with histological diagnosis of low grade advanced NEN treated unfit for systemic treatments, for one year from the start of the accrual. Endpoints and evaluation parameters:

Description of efficacy and toxicity of Temozolomide regimen in patients with advanced NENs with different primary sites unfit for systemic treatment and explored the pote ntial correlation with clinical/biological factors.

DETAILED DESCRIPTION:
Study design and trial duration This is an italian multicenter phase II trial of metronomic temozolomide in unfit patients with advanced NENs. The accrual will last 1-year and the follow up 2-year for a global 3-year period.

Objectives Primary endpoint Progression free survival (PFS).

Secondary endpoint Overall response rate (ORR) Duration of response (DOR) Overall survival (OS) Safety Quality of life (QoL)

Exploratory endpoint To evaluate O6 methylguanine DNA methyltransferase (MGMT) status in tumor tissue to validate the methods of MGMT determining and correlation with clinical outcomes

Overview on the study design Prospective analyses of consecutively NEN patients treated at Istituto Europeo di Oncologia IRCCS and participant centers between the end of 2021 and 2024 will be conducted. All patients who potentially benefit by these therapies will be proposed to participate to the study. The patient notes will then be assessed for eligibility as defined in the next section.

Treatment drug and schedule The regimen consists of oral temozolomide 60 mg once daily fasting continuously (28-day cycles)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Histologically proven diagnosis of low grade GEP-NENs (including morphology and ki67 in accordance with WHO 2019 classification), bronchial carcinoids (in accordance with the Travis classification), low grade of unknown primary sites NENs.
3. Advanced disease (unresectable locally advanced or metastatic).
4. ECOG performance status 2 and/or moderate medullary impairment (at least one of the following criteria: Hb concentration <10-8 gr/dl; WBC <3000-2000/mm3; platelets <75000-50000/mm3; neutrophil count <1500-1000/mm3); renal failure (eGFR o CrCl 30-59 ml/min - G2) and/or moderate liver failure (Child B 7-9) and/or severe comorbidities and/or > 3 prior systemic antitumor therapies (apart from SSA).

   For all the parameters other than the above mentioned criteria n° 4 consider the following criteria (that must be associated with at least one of those above): absolute neutrophil count of ≥1.5×109/L, platelet count of ≥100×109/L, haemoglobin ≥9 g/dL, serum total bilirubin <1.5 times the upper limit of normal (ULN) alanine aminotransferase (ALT), AST, or alkaline phosphatase levels ≤2.5 times the ULN (if known liver metastases ALT, AST, and ALP ≤3× the ULN), serum creatinine <1.5 times ULN or creatinine clearance ≥60 mL/min as estimated by the Cockcroft-Gault formula
5. Functioning/non functioning.
6. Morphological progressive disease (CT scan or MRI).
7. Recovery from toxicities related to any prior treatments, adequate wash-out period from previous treatments.
8. Ability to swallow pills.
9. Fertile men should agree to use effective contraceptive methods up to 6 months after the last temozolomide intake and should be informed about the possible irreversible infertility related to temozolomide intake.

Exclusion Criteria:

1. Patients pretreated with temozolomide.
2. Are Women of Child-Bearing Potential (WOCBP) and men who are able to father a child, unwilling to use adequate contraception prior to trial entry, for the duration of trial participation and for at least 28 days 2 weeks after treatment has ended. Adequate methods of contraception and Women of Child-Bearing Potential; WOCBP childbearing potential who are nursing or are pregnant or do not agree to submit to pregnancy testing required by this protocol
3. Patients that did not sign written informed consent prior to admission into the trial that is consistent with International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP) guidelines and local law
4. Knowed active hepatitis B infection (defined as presence of Hepatitis B (HepB) sAg and/or HepB DNA), active Hepatitis C (HEP C) infection (defined as presence of Hep C RNA) and/or known Human Immunodeficiency Virus (HIV) carrier.
5. Patients treated with systemic therapies (chemotherapy, interferon-alpha, somatostatin analogues, molecular target therapies) within 1 month prior to screening visit
6. Hypersensitivity to the active substance or to any of the excipients, hypersensitivity to dacarbazine (DTIC), known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 3 months before study entry, pregnant or lactating females, patients on chronic treatment with valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS). | 3 years
  PFS will be defined as the time from starting treatment to documented disease progression or death from any cause. For patients without documented progression or death at the time of analysis, PFS will be censored at the last actual visit date of tumor evaluation.

SECONDARY OUTCOMES:
Objective response rate (ORR). | 3 years
  ORR will be defined as the percentage of patients with complete responses (CR) or partial responses (PR). Patients for whom overall best response is not CR or PR, as well as patients without any post baseline tumor assessment, will be considered non responders.
Duration of response (DoR) | 3 years
  DOR will be defined as the time from the first documented objective response of PR or CR, whichever is noted earlier, to disease progression or death (if death occurs before progression is documented). DOR will be defined for responders only, i.e.
  patients with a CR or PR. DOR for patients who have not progressed or died at the time of analysis will be censored at the date of their last tumor assessment.
Overall survival (OS) | 3 years
  Overall survival (OS). OS will be defined as the time from starting treatment to death from any cause. Patients alive at the date of data cut off for analysis will be censored at the last date known to be alive.
Incidence of adverse events (AEs) | 3 years
  Incidence of adverse events (AEs), with severity determined through use of the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0); change from baseline in targeted vital signs and physical findings ; change from baseline in targeted clinical laboratory test results
Quality of life (QoL) | 3 years
  Mean changes from baseline score in patient function (physical, role, social, emotional, cognitive) and disease/treatment related symptoms by cycle, as assessed by a ll function scales and symptom items/scales of the EORTC QLQ C30, EORTC GI NET 2 and G8 test for frail elderly patients.

OTHER OUTCOMES:
Exploratory biomarker | 3 years
  O6 methylguanine DNA methyltransferase (MGMT) status will be evaluate in tumor tissue to validate the methods of MGMT determining and correlation with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Spada, MD, PhD, Principal Investigator — European Institute of Oncology (IEO), IRCCS, Milan (Italy); Nicola Fazio, MD, PhD, Study Chair — European Institute of Oncology (IEO), IRCCS, Milan (Italy)
Locations (1):
- European Institute of Oncology, IEO, IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lambrescu I, Fica S, Martins D, Spada F, Cella C, Bertani E, Rubino M, Gibelli B, Grana C, Bonomo G, Funicelli L, Ravizza D, Pisa E, Zerini D, Ungaro A, Fazio N; IEO ENETS Center of Excellence for GEP NET. Metronomic and metronomic-like therapies in neuroendocrine tumors - Rationale and clinical perspectives. Cancer Treat Rev. 2017 Apr;55:46-56. doi: 10.1016/j.ctrv.2017.02.007. Epub 2017 Feb 24. PMID 28314176
- [Result] Koumarianou A, Kaltsas G, Kulke MH, Oberg K, Strosberg JR, Spada F, Galdy S, Barberis M, Fumagalli C, Berruti A, Fazio N. Temozolomide in Advanced Neuroendocrine Neoplasms: Pharmacological and Clinical Aspects. Neuroendocrinology. 2015;101(4):274-88. doi: 10.1159/000430816. Epub 2015 Apr 29. PMID 25924937
- [Result] Weller M, Tabatabai G, Kastner B, Felsberg J, Steinbach JP, Wick A, Schnell O, Hau P, Herrlinger U, Sabel MC, Wirsching HG, Ketter R, Bahr O, Platten M, Tonn JC, Schlegel U, Marosi C, Goldbrunner R, Stupp R, Homicsko K, Pichler J, Nikkhah G, Meixensberger J, Vajkoczy P, Kollias S, Husing J, Reifenberger G, Wick W; DIRECTOR Study Group. MGMT Promoter Methylation Is a Strong Prognostic Biomarker for Benefit from Dose-Intensified Temozolomide Rechallenge in Progressive Glioblastoma: The DIRECTOR Trial. Clin Cancer Res. 2015 May 1;21(9):2057-64. doi: 10.1158/1078-0432.CCR-14-2737. Epub 2015 Feb 5. PMID 25655102
- See also: European Institute of Oncology website — https://www.ieo.it/it/PER-I-PAZIENTI/Sperimentazioni-cliniche/Sperimentazioni-cliniche/?title=MeTe&pathology=&division=&active=False
- See also: European Institute of Oncology website — https://www.ieo.it/it/PNA/Trova-Medico/?name=spada